CLINICAL TRIAL: NCT02000206
Title: Safety and Efficacy of Sedation for Flexible Fiberoptic Bronchoscopy: Comparison of Propofol/Alfentanil With Propofol/Ketamine
Brief Title: Comparison of Propofol/Alfentanil With Propofol/Ketamine
Acronym: KET-001
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Mordechai Kremer, Head of Pulmonary Institute, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RMC13ctl
Record Dates: First submitted 2013-10-23; First posted 2013-12-04 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-11

CONDITIONS: Lung Disease
Keywords: Ketamine; Alfentanil; Propofol; Oxygen saturation; Percutaneous carbon dioxide; Bronchoscopy
MeSH Terms: conditions — Lung Diseases | interventions — Propofol; Ketamine; Alfentanil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- propofol + alfentanil (Active Comparator): Patients from the Propofol / Alfentanil group will receive in addition:
  1. A loading dose of 10-15 mcg/kg Alfentanil + 0.4 mg/kg Propofol, 2 minutes prior to the beginning of the procedure.
  2. Additional boluses of Propofol (aliquots of 10-50 mg) throughout the procedure if required
  Interventions: Drug: Propofol; Drug: Alfentanil
- propofol + ketamine (Active Comparator): Patients from the Propofol / Ketamine group will receive in addition:
  1. A loading dose of 0.2-0.3 mg/kg Ketamine + 0.4 mg/kg Propofol, 2 minutes prior to the beginning of the procedure.
  2. Additional boluses of Propofol (aliquots of 10-50 mg) and/or Ketamine (aliquots of 5-25 mg) throughout the procedure if required.
  Interventions: Drug: Propofol; Drug: Ketamine

INTERVENTIONS:
Drug: Propofol
  Other Names: Diprivan
Drug: Ketamine
  Other Names: Ketalar
  Arms: propofol + ketamine
Drug: Alfentanil
  Other Names: Alfenta
  Arms: propofol + alfentanil

SUMMARY:
A prospective, randomized, patient-blinded comparison of the safety and efficacy of conscious sedation by propofol/alfentanil with propofol/ketamine in patients undergoing flexible fiberoptic bronchoscopy.

DETAILED DESCRIPTION:
The study group will include 80 patients undergoing flexible fiberoptic bronchoscopy(FFB).

Patients will be randomly assigned prior to the procedure to receive sedation by either propofol/alfentanil (PA group) or propofol/ketamine (PK group), using either the sealed envelope method or by computer randomization.

All patients will receive local anesthesia with Lidocaine 2% (total dose of 5-10 ml) that will be sprayed via the bronchoscope on the vocal cords before passage through them, as well as into the bronchial tree in order to suppress coughing.

In addition, patients from both groups will optionally receive intravenous Midazolam (up to a total dose of 0.05 mg/kg)if deemed necessary during the procedure.

Sedation will be started by 10-15 mcg/kg Alfentanil and 0.4 mg/kg Propofol, or by 0.2-0.3 mg/kg Ketamine and 0.4 mg/kg Propofol. It will be maintained by additional boluses of Propofol (aliquots of 10-50 mg) or by additional boluses of Propofol (aliquots of 10-50 mg) and/or Ketamine (aliquots of 5-25 mg).

All patients will receive supplemental oxygen via nasal cannula (2-4 L/min) before the beginning of the procedure.

Patients whose functional oxygen saturation (SpO2) prior to the beginning of the procedure will be lower than 92% while connected to a nasal cannula, will receive oxygen supplementation via a face mask.

If the SpO2 after initiation of sedation will fall below 90%, the patients' airways will be opened using a jaw-thrust maneuver or insertion of a nasal airway. Should the SpO2 remain low, the patient will receive oxygen supplementation via a face-mask.

If deemed necessary, additional safety measures will be taken by the anesthesiologist or by the performer of the bronchoscopy, such as administration of oxygen directly through the bronchoscope, assisted ventilation with an Ambu bag, and tracheal intubation.

The duration of bronchoscopy will be calculated from the administration of sedation until the flexible bronchoscope is removed from the tracheobronchial tree.

In all cases, patients will be monitored using continuous electrocardiography, pulse oximetry, and transcutaneous carbon dioxide (PtCO2, using a digital sensor placed on the patient's earlobe),and automated noninvasive blood pressure recordings every 5 minutes. All parameters will be recorded beginning from prior to connecting the patient to the nasal cannula before initiation of sedation, throughout the entire procedure and until 10 minutes after removal of the bronchoscope from the nasopharynx.

Immediately after the end of the procedure, the bronchoscopist will grade the quality of sedation (ease of performing the procedure) by Visual Analog Scale.

A questionnaire evaluating pain and discomfort by Visual Analog Scale will be completed by the patient when fully awake after the procedure.(~30 minutes after the end of the procedure).

Percutaneous carbon dioxide tension, blood oxygenation, heart rate, and blood pressure will be compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists grade I or II
* patients that will be referred to the procedure for bronchoalveolar lavage and cytologic/bacteriologic sampling, endoluminal biopsies for pathologic /bacteriologic analysis, or for regaining patency (mechanically or laser-assisted) of airways that are obstructed by secretions, tumors or foreign bodies

Exclusion Criteria:

* patient refusal or inability to provide informed consent
* American Society of Anesthesiologists grade III or higher
* allergy to study medications
* patients who have an endotracheal tube or tracheostomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-02; Primary Completion 2014-09 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Percutaneous carbon dioxide tension | Average expected time of 45 minutes
  Continuous measurements (record every 4 seconds). Throughout the duration of fiberoptic bronchoscopy - from the beginning of the procedure until 10 minutes after its termination.
oxygen saturation | Average expected time of 45 minutes.
  Continuous measurements (record every 4 seconds). Throughout the duration of fiberoptic bronchoscopy - from the beginning of the procedure until 10 minutes after its termination.
heart rate | Average expected time of 45 minutes
  Continuous measurements (record every 4 seconds). Throughout the duration of fiberoptic bronchoscopy - from the beginning of the procedure until 10 minutes after its termination.
Non-invasive blood pressure | Average expected time of 45 minutes
  Every 5 minutes. Throughout the duration of fiberoptic bronchoscopy - from the beginning of the procedure until 10 minutes after its termination

SECONDARY OUTCOMES:
Oxygen supplementation | Average expected time of 45 minutes
  Significant hypoxemia, defined as functional SpO2 of 90%, will be treated initially with a jaw thrust maneuver. If it lasts more than few seconds, a naso/oropharyngeal tube will be inserted or supplemental oxygen will be delivered via face mask at 10 L min-1.
  The percentage of patients who needed supplemental oxygen will be evaluated
Naso/oropharyngeal tube insertion | Average expected time of 45 minutes
  Significant hypoxemia, defined as functional SpO2 of 90%, will be treated initially with jaw support. If it lasts more than few seconds, a naso/oropharyngeal tube will be inserted or supplemental oxygen will be delivered via face mask at 10 L min-1
  The percentage of patients who needed Naso/oropharyngeal tube insertion will be evaluated
A questionnaire evaluating pain and discomfort | Ca. 30 minutes after the end of the procedure (average expected time of 60 minutes)
  A questionnaire evaluating pain and discomfort by Visual Analog Scale will be completed by the patient when awake after the procedure.(~30 minutes after the end of the procedure)
A questionnaire evaluating the quality of sedation | Immediately after end of procedure (average expected time of 30 minutes)
  A questionnaire evaluating the quality of sedation and the ease of performing the procedure by Visual Analog Scale will be completed by the bronchoscopist immediately after the procedure.
Total propofol dosage | Average expected time of 30 minutes
  The total amount of propofol used throughout the procedure will be calculated.
Time to full awakening and orientation | Anticipated to be in the range of 1-30 minutes after the end of the procedure
  Time from termination of the procedure to full awakening and orientation
Time to discharge | Average expected time of 60 minutes. Anticipated to be in the range of 45-120 minutes after the end of fiberoptic bronchoscopy
  The time from the termination of the procedure until the patient is discharged from the recovery unit will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Mordechai R Kramer, MD, Study Director — Rabin Medical Center
Locations (1):
- Pulmonary Institute, Rabin Medical Center, Beilinson Hospital, Petah Tikva, Israel

REFERENCES:
- [Background] Stolz D, Chhajed PN, Leuppi JD, Brutsche M, Pflimlin E, Tamm M. Cough suppression during flexible bronchoscopy using combined sedation with midazolam and hydrocodone: a randomised, double blind, placebo controlled trial. Thorax. 2004 Sep;59(9):773-6. doi: 10.1136/thx.2003.019836. PMID 15333854
- [Background] British Thoracic Society Bronchoscopy Guidelines Committee, a Subcommittee of Standards of Care Committee of British Thoracic Society. British Thoracic Society guidelines on diagnostic flexible bronchoscopy. Thorax. 2001 Mar;56 Suppl 1(Suppl 1):i1-21. doi: 10.1136/thorax.56.suppl_1.i1. No abstract available. PMID 11158709
- [Background] Gonzalez R, De-La-Rosa-Ramirez I, Maldonado-Hernandez A, Dominguez-Cherit G. Should patients undergoing a bronchoscopy be sedated? Acta Anaesthesiol Scand. 2003 Apr;47(4):411-5. doi: 10.1034/j.1399-6576.2003.00061.x. PMID 12694138
- [Background] Fox BD, Krylov Y, Leon P, Ben-Zvi I, Peled N, Shitrit D, Kramer MR. Benzodiazepine and opioid sedation attenuate the sympathetic response to fiberoptic bronchoscopy. Prophylactic labetalol gave no additional benefit. Results of a randomized double-blind placebo-controlled study. Respir Med. 2008 Jul;102(7):978-83. doi: 10.1016/j.rmed.2008.02.011. Epub 2008 Apr 3. PMID 18394874
- [Background] Putinati S, Ballerin L, Corbetta L, Trevisani L, Potena A. Patient satisfaction with conscious sedation for bronchoscopy. Chest. 1999 May;115(5):1437-40. doi: 10.1378/chest.115.5.1437. PMID 10334165
- [Background] Stolz D, Kurer G, Meyer A, Chhajed PN, Pflimlin E, Strobel W, Tamm M. Propofol versus combined sedation in flexible bronchoscopy: a randomised non-inferiority trial. Eur Respir J. 2009 Nov;34(5):1024-30. doi: 10.1183/09031936.00180808. Epub 2009 Apr 22. PMID 19386684
- [Background] Clark G, Licker M, Younossian AB, Soccal PM, Frey JG, Rochat T, Diaper J, Bridevaux PO, Tschopp JM. Titrated sedation with propofol or midazolam for flexible bronchoscopy: a randomised trial. Eur Respir J. 2009 Dec;34(6):1277-83. doi: 10.1183/09031936.00142108. Epub 2009 May 14. PMID 19443532
- [Background] Crawford M, Pollock J, Anderson K, Glavin RJ, MacIntyre D, Vernon D. Comparison of midazolam with propofol for sedation in outpatient bronchoscopy. Br J Anaesth. 1993 Apr;70(4):419-22. doi: 10.1093/bja/70.4.419. PMID 8499201
- [Background] White PF, Way WL, Trevor AJ. Ketamine--its pharmacology and therapeutic uses. Anesthesiology. 1982 Feb;56(2):119-36. doi: 10.1097/00000542-198202000-00007. No abstract available. PMID 6892475
- [Background] Berkenbosch JW, Graff GR, Stark JM. Safety and efficacy of ketamine sedation for infant flexible fiberoptic bronchoscopy. Chest. 2004 Mar;125(3):1132-7. doi: 10.1378/chest.125.3.1132. PMID 15006978
- [Background] Slonim AD, Ognibene FP. Amnestic agents in pediatric bronchoscopy. Chest. 1999 Dec;116(6):1802-8. doi: 10.1378/chest.116.6.1802. PMID 10593809
- [Background] Hwang J, Jeon Y, Park HP, Lim YJ, Oh YS. Comparison of alfetanil and ketamine in combination with propofol for patient-controlled sedation during fiberoptic bronchoscopy. Acta Anaesthesiol Scand. 2005 Oct;49(9):1334-8. doi: 10.1111/j.1399-6576.2005.00842.x. PMID 16146472